CLINICAL TRIAL: NCT00003291
Title: Molecular Genetic Lesions and Clinical Outcome in Pediatric ALL Patients
Brief Title: Molecular Genetic Lesions and Clinical Outcomes in Children With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: B969; COG-B969 (Other: Children's Oncology Group); CCG-B969 (Other: Children's Cancer Group); CDR0000066224 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cytogenetic Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: mutation analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: The identification of gene mutations may allow doctors to better determine the prognosis of children with acute lymphoblastic leukemia.

PURPOSE: This clinical trial is studying gene mutations to see if they are related to prognosis of cancer in children with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the prognostic significance of deletion of the p16 (MTS1, CDKN21) gene in children with acute lymphoblastic leukemia.
* Attempt to correlate the incidence of specific, nonrandom combinations of molecular genetic lesions with clinical outcome in these patients.

OUTLINE: Patients are stratified by risk (standard vs high).

Bone marrow specimens from patients enrolled in CCG-1922, CCG-1882, or CCG-1901 are analyzed for the following genetic lesions: p16 deletion, p14 deletion, and p15 deletion.

Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

Patients are followed for at least 3 years.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia (ALL)
* Meets criteria for 1 of the following:

  * Standard risk, as defined by the following:

    * 1 to 10 years old at diagnosis
    * WBC less than 50,000/mm^3
  * High risk, as defined by the following:

    * Less than 1 year old or over 10 years old at diagnosis
    * WBC greater than 50,000/mm^3
* Enrolled on CCG-1922 (standard-risk ALL) or CCG-1882 or CCG-1901 (high-risk ALL)

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 1998-03; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula R. Kees, PhD, Study Chair — Telethon Institute for Child Health Research
Locations (1):
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia